CLINICAL TRIAL: NCT05019053
Title: Acceptability/Feasibility of COVID-19 Intervention of a Virtual Group Intervention for COVID-19 Distress
Brief Title: Acceptability/Feasibility of COVID-19 Intervention
Acronym: COPING CREW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Nicholas Allan, Assistant Professor of Clinical Psychology, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAKER_Coping Crew Intervention
Record Dates: First submitted 2021-07-29; First posted 2021-08-24 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Social Isolation; Emotional Disorder
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coping Crew Intervention (Experimental): Interested participants who meet the screening criteria will be assigned to receive COPING CREW. First, following informed consent, eligible participants will complete a baseline assessment appointment in the week prior to the group beginning. During the baseline appointment, participants will provide informed consent, be instructed in the use of Microsoft Teams, complete a battery of self-report measures, be given a semi-structured diagnostic interview, and follow instructions to install a mobile app that will be used to track their mood and homework. Then, 4 groups of COPING CREW, with 6 participants per group, will be run. Participants will complete four weekly 60-minute virtual intervention sessions followed by a booster session two weeks later. Participants will complete daily surveys and homework assignments on their mobile devices. Links to follow-up surveys will be sent to participants at 1- and 3-month follow-ups.
  Interventions: Behavioral: Coping Crew

INTERVENTIONS:
Behavioral: Coping Crew — Coping Crew consists of five 60-minute virtual intervention sessions coinciding with five weeks of EMI. Participants will receive psychoeducation, challenge cognitive biases or mythbust, and participate in behavioral exposure and behavioral experiments. An EMI component of this treatment will be included for the purpose of treatment monitoring and homework tracking. Participation in this EMI component involves the daily report of levels of anxiety, depression, stress, and loneliness. When participants endorse elevated levels on any of these constructs, they will receive a targeted message reminding them of the topics covered in COPING CREW. One month after the intervention session, COPING CREW participants will complete follow-up questionnaires and interview. Participants will also participate in a feedback session 3 months after the intervention.

SUMMARY:
The coronavirus (COVID-19) pandemic is a significant psychological stressor that threatens the onset of a mental health crisis in the US. Fear and anxiety about COVID-19 and its economic impact, as well as loneliness due to the required social isolation, are driving the mental health impacts of COVID-19; in a recent Kaiser Family Foundation poll, 45% of respondents reported that the coronavirus has had a negative impact on their mental health. This is reflected in Southeastern Ohio. In data that the investigators collected from 317 Ohio University faculty, staff, and students from late May to early June, 39% reported moderate-to-severe levels of anxiety, 41% reported moderate-to-severe levels of depression and 57% reported the COVID-19 outbreak was impacting their sense of social connection much or very much. Despite the significant community need for accessible and affordable care, there are currently no evidence-based interventions for individuals coping poorly with coronavirus-related distress. The investigators have developed a virtual group-based intervention targeting cognitive biases that amplify the experience of stress and anxiety (i.e., amplifying cognitions; Coping with Coronavirus-Related Emotion and Worry [COPING CREW]). The next step in developing this intervention in a scientifically rigorous manner is to refine the manual and procedures and conduct a pilot test of the intervention.

DETAILED DESCRIPTION:
There is a coming mental health crisis in response to the COVID-19 pandemic. Already, rates of depression, anxiety, and suicide are elevated in response to the pandemic. A recent study of more than 5,400 people in the US found prevalence rates of anxiety and depression in June of 2020 were 3-4 times higher than these rates in June of 2019. In this same study, 41% of respondents in June 2020 reported experiencing an adverse mental or behavioral health condition, including 13% who endorsed using substances to cope with stress or emotions and 11% who reported seriously contemplating suicide in the prior 30 days. Thus, heightened anxiety, stress, and depression will likely continue to lead to increases in self-harm and maladaptive substance use if left unchecked.

It is crucial that empirically validated psychotherapies be developed to meet these needs. These treatments must address how common barriers to treatment, including time, cost, transportation, and stigma about mental health may be exacerbated by the pandemic. The investigators developed a brief, virtual group-based intervention, framed as educational, Coping with Coronavirus-Related Emotions and Worries (COPING CREW), to address these barriers. This intervention was developed over the summer by Drs. Allan, Suhr, and Austin, working with two graduate student research assistants for administration by clinical psychology graduate student therapists as part of their practicum experience at the Ohio University Psychology and Social Work Clinic (PSWC). A benefit of this approach, therefore, is that this intervention is highly scalable.

Theoretical models posit the short- and long-term stressors experienced during the pandemic exacerbate the experience of negative emotions an individual is already predisposed to experience. That is, people who are already experiencing mental health issues are going to experience more severe issues and people who may not already be experiencing mental health issues are more likely to develop mental health issues during the pandemic. Cognitive risk factors (i.e., amplifying cognitions) such as anxiety sensitivity (fear of anxiety sensations), intolerance of uncertainty (fear of the unknown), and loneliness (the subjective feeling of isolation) increase the experience of negative emotions as well as the likelihood of unhealthy coping behavior such as increased alcohol consumption or self-harm.

Anxiety sensitivity, intolerance of uncertainty, and loneliness can be reduced through brief interventions applying cognitive-behavioral therapy principles. Reductions in these constructs lead to later reductions in anxiety, depression, and suicide. Targeting these risk factors appears critical to address distress due to COVID-19. In 317 Ohio University faculty, staff, and students, anxiety sensitivity, intolerance of uncertainty, and loneliness accounted for 63%-75% of the variance in ratings of anxiety, depression, and suicidality as well as 49% of COVID-related disability. These findings highlight the prominent role these risk factors play in the distress many individuals are experiencing due to COVID-19. The investigators have developed a virtual group-based intervention targeting risk factors that amplify the experience of emotional distress; the next steps in developing a scientifically rigorous intervention that can be disseminated broadly is to develop and pilot test this intervention.

The goals specific to this project are to 1) engage stakeholders in the design of a brief group-based treatment to improve COPING CREW and 2) to conduct a Stage I pilot trial through evaluating the acceptability and feasibility of COPING CREW.

Aim 1: Refine a prototype for COPING CREW by working virtually with a community partner stakeholder advisory group (SAG) as well as participants receiving the intervention. The investigators will develop a SAG comprising one participant from each community partner. The investigators will meet with the SAG at least three times during the 1-year project. Meetings will occur prior to starting COPING CREW groups, after running the first two groups, and after all four groups have been completed. The investigators anticipate that building a strong relationship with this SAG will increase treatment relevance to clientele, treatment engagement, and treatment dissemination. In turn, this will enhance the durable impacts and sustainability of COPING CREW. In addition to SAGs, the investigators will also utilize a systematic approach to engage with participant stakeholders by asking for feedback about the intervention (the Exit Interview). The investigators have used these intervention modules separately a number of times but have yet to examine these modules as part of the same intervention. Thus, participants will provide important information on how to tailor the intervention, including the order of the components, the amount of homework specific to each component, and the length of time before the booster session to best meet their needs. Although the investigators are confident that COPING CREW will largely be viewed as acceptable, it can be modified to increase acceptability by effective engagement with community partners. Solicitation of feedback will occur via two mechanisms. First, information related to adaptation will be obtained from quantitative and qualitative feedback during the intervention. Second, information related to adaptation and engagement will also be collected in separate, focused feedback sessions with COPING CREW participants.

Aim 2: Examine acceptability and feasibility of COPING CREW, delivered virtually. A pilot one arm trial will be conducted, delivering the intervention to 24 participants across 4 groups.

H1: It is hypothesized that the intervention will demonstrate high acceptability and feasibility (as measured by completion rates and favorable ratings of satisfaction) across intervention modules and components within sessions. Components will include psychoeducation, challenging cognitive biases or mythbusting, behavioral exposure, behavioral experiments, and ecological momentary intervention (EMI) for treatment monitoring and homework tracking.

ELIGIBILITY:
Inclusion Criteria:

* Elevated anxiety sensitivity (i.e., a score greater than 1 standard deviation above the mean on the Anxiety Sensitivity Index-3; Taylor et al., 2007)
* Elevated Intolerance of uncertainty (i.e., a score greater than 1 standard deviation above the mean on the Intolerance of Uncertainty Scale - Short Form; Carleton et al., 2007)
* Elevated loneliness (i.e., a score greater than 1 standard deviation above the mean on the NIH Toolbox Loneliness Scale; Cyranowski et al., 2013)
* Access to a device with internet connection

Exclusion Criteria:

* Participants who have previously received other FEAR Lab interventions or participated in a focus group related to that intervention (20-X-184; 20-X-204) will be excluded due to the overlap of intervention material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the intervention as assessed by Client Satisfaction Questionnaire-8 | Immediately after the intervention
  The Client Satisfaction Questionnaire-8 is a 8-item self-report scale that assesses client satisfaction with a particular intervention/program. The Client Satisfaction Questionnaire-8 is completed by rating satisfaction with services on a 1-4 Likert-type scale. Possible total scores range from 8 to 32. Greater satisfaction is indicated by higher scores.
Feasibility of service as assessed by response rates for the Ecological Momentary Assessment/Ecological Momentary Intervention component of the intervention | 5-week EMA/EMI, During the Intervention (Weeks 1-5)
  Feasibility will also be determined based on response rates for Ecological Momentary Assessment/Ecological Momentary Intervention. If 80% of participants respond to 80% of the EMA prompts, this will be considered a feasible means of service delivery.

SECONDARY OUTCOMES:
COVID-19 Impact Battery - Behavior | Baseline, pre-intervention
  This 12-item scale was created to measure behavioral patterns in response to the COVID-19 outbreak. Participants responded to this scale by rating the extent to which they "have engaged in the following behaviors in response to COVID-19" using a five-point scale (from 0 = "Not at all" to 4 = "Very much"). Each of the potential behaviors listed in this scale (e.g., "Using hand sanitizer") were rated by participants. Possible total scores range from 0 to 48. A higher rate of engagement in the listed behaviors is indicated by a higher score.
COVID-19 Impact Battery - Behavior | Immediately after the intervention
  This 12-item scale was created to measure behavioral patterns in response to the COVID-19 outbreak. Participants responded to this scale by rating the extent to which they "have engaged in the following behaviors in response to COVID-19" using a five-point scale (from 0 = "Not at all" to 4 = "Very much"). Each of the potential behaviors listed in this scale (e.g., "Using hand sanitizer") were rated by participants. Possible total scores range from 0 to 48. A higher rate of engagement in the listed behaviors is indicated by a higher score.
COVID-19 Impact Battery - Behavior | Follow-Up, 1 month after the intervention
  This 12-item scale was created to measure behavioral patterns in response to the COVID-19 outbreak. Participants responded to this scale by rating the extent to which they "have engaged in the following behaviors in response to COVID-19" using a five-point scale (from 0 = "Not at all" to 4 = "Very much"). Each of the potential behaviors listed in this scale (e.g., "Using hand sanitizer") were rated by participants. Possible total scores range from 0 to 48. A higher rate of engagement in the listed behaviors is indicated by a higher score.
COVID-19 Impact Battery - Behavior | Follow-Up, 3 months after the intervention
  This 12-item scale was created to measure behavioral patterns in response to the COVID-19 outbreak. Participants responded to this scale by rating the extent to which they "have engaged in the following behaviors in response to COVID-19" using a five-point scale (from 0 = "Not at all" to 4 = "Very much"). Each of the potential behaviors listed in this scale (e.g., "Using hand sanitizer") were rated by participants. Possible total scores range from 0 to 48. A higher rate of engagement in the listed behaviors is indicated by a higher score.
COVID-19 Impact Battery - Worry | Baseline, pre-intervention
  This 11-item scale was created to measure worry and distress in response to the outbreak of COVID-19. The items on this measure use a five-point scale (from 0 = "Not at all" to 4 = "Very Much"). Participants used this scale to rate each item (e.g., "I worry that I will lose my employment") based on the degree to which it has caused distress. Possible total scores range from 0 to 44. Greater worry and distress is indicated by higher scores.
COVID-19 Impact Battery - Worry | Immediately after the intervention
  This 11-item scale was created to measure worry and distress in response to the outbreak of COVID-19. The items on this measure use a five-point scale (from 0 = "Not at all" to 4 = "Very Much"). Participants used this scale to rate each item (e.g., "I worry that I will lose my employment") based on the degree to which it has caused distress. Possible total scores range from 0 to 44. Greater worry and distress is indicated by higher scores.
COVID-19 Impact Battery - Worry | Follow-Up, 1 month after the intervention
  This 11-item scale was created to measure worry and distress in response to the outbreak of COVID-19. The items on this measure use a five-point scale (from 0 = "Not at all" to 4 = "Very Much"). Participants used this scale to rate each item (e.g., "I worry that I will lose my employment") based on the degree to which it has caused distress. Possible total scores range from 0 to 44. Greater worry and distress is indicated by higher scores.
COVID-19 Impact Battery - Worry | Follow-Up, 3 months after the intervention
  This 11-item scale was created to measure worry and distress in response to the outbreak of COVID-19. The items on this measure use a five-point scale (from 0 = "Not at all" to 4 = "Very Much"). Participants used this scale to rate each item (e.g., "I worry that I will lose my employment") based on the degree to which it has caused distress. Possible total scores range from 0 to 44. Greater worry and distress is indicated by higher scores.
COVID-19 Impact Battery - Disability | Baseline, pre-intervention
  This 7-item scale was created to measure the presence of difficulties in response to the outbreak of COVID-19. Participants were asked to rate difficulties on a five-point scale from 0 ("None") to 4 ("Extreme or cannot do"). Participants used this scale to rate the degree of difficulties experienced in the preceding 30 days because of the COVID-19 outbreak. Possible total scores range from 0 to 28. A greater rate of disability is indicated by a higher score.
COVID-19 Impact Battery - Disability | Immediately after the intervention
  This 7-item scale was created to measure the presence of difficulties in response to the outbreak of COVID-19. Participants were asked to rate difficulties on a five-point scale from 0 ("None") to 4 ("Extreme or cannot do"). Participants used this scale to rate the degree of difficulties experienced in the preceding 30 days because of the COVID-19 outbreak. Possible total scores range from 0 to 28. A greater rate of disability is indicated by a higher score.
COVID-19 Impact Battery - Disability | Follow-Up, 1 month after the intervention
  This 7-item scale was created to measure the presence of difficulties in response to the outbreak of COVID-19. Participants were asked to rate difficulties on a five-point scale from 0 ("None") to 4 ("Extreme or cannot do"). Participants used this scale to rate the degree of difficulties experienced in the preceding 30 days because of the COVID-19 outbreak. Possible total scores range from 0 to 28. A greater rate of disability is indicated by a higher score.
COVID-19 Impact Battery - Disability | Follow-Up, 3 months after the intervention
  This 7-item scale was created to measure the presence of difficulties in response to the outbreak of COVID-19. Participants were asked to rate difficulties on a five-point scale from 0 ("None") to 4 ("Extreme or cannot do"). Participants used this scale to rate the degree of difficulties experienced in the preceding 30 days because of the COVID-19 outbreak. Possible total scores range from 0 to 28. A greater rate of disability is indicated by a higher score.
COVID-19 Items | Baseline, pre-intervention
  Investigator-created questions assessing demographic information related to the COVID-19 pandemic will be administered.
Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale | Baseline, pre-intervention
  The PROMIS Anxiety scale is an 8-item scale that measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater anxiety is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale | During the Intervention (Weeks 1-5)
  The PROMIS Anxiety scale is an 8-item scale that measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater anxiety is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale | Immediately after the intervention
  The PROMIS Anxiety scale is an 8-item scale that measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater anxiety is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale | Follow-Up, 1 month after the intervention
  The PROMIS Anxiety scale is an 8-item scale that measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater anxiety is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety scale | Follow-Up, 3 months after the intervention
  The PROMIS Anxiety scale is an 8-item scale that measures anxiety broadly, including items to assess fear, anxious misery, hyperarousal, and somatic symptoms. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater anxiety is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale | Baseline, pre-intervention
  The PROMIS Depression scale is an 8-item scale that measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater depression is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale | During the Intervention (Weeks 1-5)
  The PROMIS Depression scale is an 8-item scale that measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater depression is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale | Immediately after the intervention
  The PROMIS Depression scale is an 8-item scale that measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater depression is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale | Follow-Up, 1 month after the intervention
  The PROMIS Depression scale is an 8-item scale that measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater depression is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) depression scale | Follow-Up, 3 months after the intervention
  The PROMIS Depression scale is an 8-item scale that measures depression. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater depression is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) stress scale | Baseline, pre-intervention
  The PROMIS Psychological Stress scale is an 8-item scale that measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater stress is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) stress scale | During the Intervention (Weeks 1-5)
  The PROMIS Psychological Stress scale is an 8-item scale that measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater stress is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) stress scale | Immediately after the intervention
  The PROMIS Psychological Stress scale is an 8-item scale that measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater stress is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) stress scale | Follow-Up, 1 month after the intervention
  The PROMIS Psychological Stress scale is an 8-item scale that measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater stress is indicated by higher scores.
Patient-Reported Outcomes Measurement Information System (PROMIS) stress scale | Follow-Up, 3 months after the intervention
  The PROMIS Psychological Stress scale is an 8-item scale that measures feelings about self and the world in the context of challenges. Items are on a 5-point scale from 1 (Never) to 5 (Always). Possible total scores range from 8 to 40. Greater stress is indicated by higher scores.
Anxiety Sensitivity Index 3 (ASI-3) | Baseline, pre-intervention
  18-item self-report measure of anxiety sensitivity. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the previous ASIs provided. The ASI-3 will be utilized to assess level of overall anxiety sensitivity. Participants are asked to rate the degree to which anxiety symptoms are distressing on a five-point scale from 0 ("Very Little") to 4 ("Very Much"). Possible total scores range from 0 to 72. Greater distress is indicated by higher scores.
Anxiety Sensitivity Index 3 (ASI-3) | During the Intervention (Weeks 1-5)
  18-item self-report measure of anxiety sensitivity. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the previous ASIs provided. The ASI-3 will be utilized to assess level of overall anxiety sensitivity. Participants are asked to rate the degree to which anxiety symptoms are distressing on a five-point scale from 0 ("Very Little") to 4 ("Very Much"). Possible total scores range from 0 to 72. Greater distress is indicated by higher scores.
Anxiety Sensitivity Index 3 (ASI-3) | Immediately after the intervention
  18-item self-report measure of anxiety sensitivity. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the previous ASIs provided. The ASI-3 will be utilized to assess level of overall anxiety sensitivity. Participants are asked to rate the degree to which anxiety symptoms are distressing on a five-point scale from 0 ("Very Little") to 4 ("Very Much"). Possible total scores range from 0 to 72. Greater distress is indicated by higher scores.
Anxiety Sensitivity Index 3 (ASI-3) | Follow-Up, 1 month after the intervention
  18-item self-report measure of anxiety sensitivity. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the previous ASIs provided. The ASI-3 will be utilized to assess level of overall anxiety sensitivity. Participants are asked to rate the degree to which anxiety symptoms are distressing on a five-point scale from 0 ("Very Little") to 4 ("Very Much"). Possible total scores range from 0 to 72. Greater distress is indicated by higher scores.
Anxiety Sensitivity Index 3 (ASI-3) | Follow-Up, 3 months after the intervention
  18-item self-report measure of anxiety sensitivity. This scale was developed to provide a more stable measure of the three most widely recognized AS subfactors (cognitive, social and physical concerns) than the previous ASIs provided. The ASI-3 will be utilized to assess level of overall anxiety sensitivity. Participants are asked to rate the degree to which anxiety symptoms are distressing on a five-point scale from 0 ("Very Little") to 4 ("Very Much"). Possible total scores range from 0 to 72. Greater distress is indicated by higher scores.
Intolerance of Uncertainty-12 | Baseline, pre-intervention
  This scale is a 12-item scale for measuring trait Intolerance of Uncertainty. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future. This scale uses a five-point, Likert-type scale ranging from 1 ("Not at all characteristic of me") to 5 ("Entirely characteristic of me"). Possible total scores range from 12 to 60. Greater uncertainty is indicated by higher scores.
Intolerance of Uncertainty-12 | During the Intervention (Weeks 1-5)
  This scale is a 12-item scale for measuring trait Intolerance of Uncertainty. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future. This scale uses a five-point, Likert-type scale ranging from 1 ("Not at all characteristic of me") to 5 ("Entirely characteristic of me"). Possible total scores range from 12 to 60. Greater uncertainty is indicated by higher scores.
Intolerance of Uncertainty-12 | Immediately after the intervention
  This scale is a 12-item scale for measuring trait Intolerance of Uncertainty. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future. This scale uses a five-point, Likert-type scale ranging from 1 ("Not at all characteristic of me") to 5 ("Entirely characteristic of me"). Possible total scores range from 12 to 60. Greater uncertainty is indicated by higher scores.
Intolerance of Uncertainty-12 | Follow-Up, 1 month after the intervention
  This scale is a 12-item scale for measuring trait Intolerance of Uncertainty. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future. This scale uses a five-point, Likert-type scale ranging from 1 ("Not at all characteristic of me") to 5 ("Entirely characteristic of me"). Possible total scores range from 12 to 60. Greater uncertainty is indicated by higher scores.
Intolerance of Uncertainty-12 | Follow-Up, 3 months after the intervention
  This scale is a 12-item scale for measuring trait Intolerance of Uncertainty. it is used for assessing the degree to which individuals are able to tolerate the uncertainty of ambiguous situations, the cognitive and behavioral responses to uncertainty, perceived implications of uncertainty, and attempts to control the future. This scale uses a five-point, Likert-type scale ranging from 1 ("Not at all characteristic of me") to 5 ("Entirely characteristic of me"). Possible total scores range from 12 to 60. Greater uncertainty is indicated by higher scores.
Insomnia Severity Index (ISI) | Baseline, pre-intervention
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four. Possible total scores range from 0 to 28. Higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Insomnia Severity Index (ISI) | Immediately after the intervention
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four. Possible total scores range from 0 to 28. Higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Insomnia Severity Index (ISI) | Follow-Up, 1 month after the intervention
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four. Possible total scores range from 0 to 28. Higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Insomnia Severity Index (ISI) | Follow-Up, 3 months after the intervention
  The ISI is a seven-item self-report questionnaire designed to assess sleep difficulties (i.e., falling asleep, staying asleep, waking too early), satisfaction/dissatisfaction with sleep patterns, and/or interference with daily functioning. Participants will be asked to rate each item using a five-point Likert-type scale ranging from zero to four. Possible total scores range from 0 to 28. Higher scores reflecting more severe sleep problems and greater dissatisfaction with sleep.
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Baseline, pre-intervention
  The DSI-SS is a 4-item measure of symptoms of suicide. The DSI-SS was designed to be a brief screening measure for suicide risk, and has well established cut points for clinical and research utility. Participants are asked to rate each item using a scale that ranges from 0 to 3 (total score range 0-12), with higher scores reflecting greater severity of suicidal ideation.
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Immediately after the intervention
  The DSI-SS is a 4-item measure of symptoms of suicide. The DSI-SS was designed to be a brief screening measure for suicide risk, and has well established cut points for clinical and research utility. Participants are asked to rate each item using a scale that ranges from 0 to 3 (total score range 0-12), with higher scores reflecting greater severity of suicidal ideation.
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Follow-Up, 1 month after the intervention
  The DSI-SS is a 4-item measure of symptoms of suicide. The DSI-SS was designed to be a brief screening measure for suicide risk, and has well established cut points for clinical and research utility. Participants are asked to rate each item using a scale that ranges from 0 to 3 (total score range 0-12), with higher scores reflecting greater severity of suicidal ideation.
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Follow-Up, 3 months after the intervention
  The DSI-SS is a 4-item measure of symptoms of suicide. The DSI-SS was designed to be a brief screening measure for suicide risk, and has well established cut points for clinical and research utility. Participants are asked to rate each item using a scale that ranges from 0 to 3 (total score range 0-12), with higher scores reflecting greater severity of suicidal ideation.
Alcohol Use Disorder Identification Test (AUDIT) | Baseline, pre-intervention
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior. For items 1-8, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 9 and 10, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 40. Greater alcohol consumption, drinking behavior, and alcohol-related problems is indicated by higher scores.
Alcohol Use Disorder Identification Test (AUDIT) | Immediately after the intervention
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior. For items 1-8, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 9 and 10, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 40. Greater alcohol consumption, drinking behavior, and alcohol-related problems is indicated by higher scores.
Alcohol Use Disorder Identification Test (AUDIT) | Follow-Up, 1 month after the intervention
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior. For items 1-8, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 9 and 10, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 40. Greater alcohol consumption, drinking behavior, and alcohol-related problems is indicated by higher scores.
Alcohol Use Disorder Identification Test (AUDIT) | Follow-Up, 3 months after the intervention
  The AUDIT is a 10-item questionnaire that assesses alcohol consumption, drinking behavior, and alcohol-related problems. The AUDIT will be administered to assess drinking behavior. For items 1-8, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 9 and 10, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 40. Greater alcohol consumption, drinking behavior, and alcohol-related problems is indicated by higher scores.
Drug Use Disorders Identification Test (DUDIT) | Baseline, pre-intervention
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior. For items 1-9, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 10 and 11, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 44. Greater drug consumption, drug use behavior, and drug-related problems is indicated by higher scores.
Drug Use Disorders Identification Test (DUDIT) | Immediately after the intervention
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior. For items 1-9, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 10 and 11, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 44. Greater drug consumption, drug use behavior, and drug-related problems is indicated by higher scores.
Drug Use Disorders Identification Test (DUDIT) | Follow-Up, 1 month after the intervention
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior. For items 1-9, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 10 and 11, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 44. Greater drug consumption, drug use behavior, and drug-related problems is indicated by higher scores.
Drug Use Disorders Identification Test (DUDIT) | Follow-Up, 3 months after the intervention
  The DUDIT is an 11-item questionnaire that assesses drug consumption, drug use behavior, and drug-related problems. The DUDIT will be administered to assess drug use behavior. For items 1-9, participants are asked to rate each item using a scale that ranges from 0 to 4. For items 10 and 11, participants are asked to choose from possible responses of 0, 2 and 4. Possible total scores range from 0 to 44. Greater drug consumption, drug use behavior, and drug-related problems is indicated by higher scores.
Fear of Arousal Questionnaire (FAQ) | Baseline, pre-intervention
  The FAQ is a 12-item self-report measure of fear of arousal. Fear of arousal is defined as the fear of the physiological responses that are typical of anxiety (e.g., racing thoughts, racing heart, or throat tightening). The measure asks participants to rate each item on a 1 to 5 scale with 1 corresponding to no anxiety and 5 corresponding to extreme anxiety. Possible total scores range from 12 to 60. Greater fear of arousal is indicated by higher scores.
Fear of Arousal Questionnaire (FAQ) | Immediately after the intervention
  The FAQ is a 12-item self-report measure of fear of arousal. Fear of arousal is defined as the fear of the physiological responses that are typical of anxiety (e.g., racing thoughts, racing heart, or throat tightening). The measure asks participants to rate each item on a 1 to 5 scale with 1 corresponding to no anxiety and 5 corresponding to extreme anxiety. Possible total scores range from 12 to 60. Greater fear of arousal is indicated by higher scores.
Fear of Arousal Questionnaire (FAQ) | Follow-Up, 1 month after the intervention
  The FAQ is a 12-item self-report measure of fear of arousal. Fear of arousal is defined as the fear of the physiological responses that are typical of anxiety (e.g., racing thoughts, racing heart, or throat tightening). The measure asks participants to rate each item on a 1 to 5 scale with 1 corresponding to no anxiety and 5 corresponding to extreme anxiety. Possible total scores range from 12 to 60. Greater fear of arousal is indicated by higher scores.
Fear of Arousal Questionnaire (FAQ) | Follow-Up, 3 months after the intervention
  The FAQ is a 12-item self-report measure of fear of arousal. Fear of arousal is defined as the fear of the physiological responses that are typical of anxiety (e.g., racing thoughts, racing heart, or throat tightening). The measure asks participants to rate each item on a 1 to 5 scale with 1 corresponding to no anxiety and 5 corresponding to extreme anxiety. Possible total scores range from 12 to 60. Greater fear of arousal is indicated by higher scores.
National Institutes of Health (NIH) Toolbox Loneliness Scale | Baseline, pre-intervention
  The NIH Toolbox Loneliness Scale is a 5-item scale belonging to the NIH Toolbox Adult Social Relationship Scales. This brief scale was developed to measure perceived loneliness, or the perception that one is lonely or socially isolated from others. The measure asks participants to rate each item on a 1 ("Never") to 5 ("Always") scale. Possible total scores range from 5 to 25. Greater loneliness is indicated by higher scores.
National Institutes of Health (NIH) Toolbox Loneliness Scale | During the Intervention (Weeks 1-5)
  The NIH Toolbox Loneliness Scale is a 5-item scale belonging to the NIH Toolbox Adult Social Relationship Scales. This brief scale was developed to measure perceived loneliness, or the perception that one is lonely or socially isolated from others. The measure asks participants to rate each item on a 1 ("Never") to 5 ("Always") scale. Possible total scores range from 5 to 25. Greater loneliness is indicated by higher scores.
National Institutes of Health (NIH) Toolbox Loneliness Scale | Immediately after the intervention
  The NIH Toolbox Loneliness Scale is a 5-item scale belonging to the NIH Toolbox Adult Social Relationship Scales. This brief scale was developed to measure perceived loneliness, or the perception that one is lonely or socially isolated from others. The measure asks participants to rate each item on a 1 ("Never") to 5 ("Always") scale. Possible total scores range from 5 to 25. Greater loneliness is indicated by higher scores.
National Institutes of Health (NIH) Toolbox Loneliness Scale | Follow-Up, 1 month after the intervention
  The NIH Toolbox Loneliness Scale is a 5-item scale belonging to the NIH Toolbox Adult Social Relationship Scales. This brief scale was developed to measure perceived loneliness, or the perception that one is lonely or socially isolated from others. The measure asks participants to rate each item on a 1 ("Never") to 5 ("Always") scale. Possible total scores range from 5 to 25. Greater loneliness is indicated by higher scores.
National Institutes of Health (NIH) Toolbox Loneliness Scale | Follow-Up, 3 months after the intervention
  The NIH Toolbox Loneliness Scale is a 5-item scale belonging to the NIH Toolbox Adult Social Relationship Scales. This brief scale was developed to measure perceived loneliness, or the perception that one is lonely or socially isolated from others. The measure asks participants to rate each item on a 1 ("Never") to 5 ("Always") scale. Possible total scores range from 5 to 25. Greater loneliness is indicated by higher scores.
Exit Interview | Immediately after the intervention
  Participants will provide information on how to tailor the intervention, including the order of the components, the amount of homework specific to each component, and the length of time before the booster session to best meet their needs. They will provide this information in a focused feedback session in which they will respond to an investigator-created semi-structured interview.
Ecological Momentary Assessment (EMA) questions | During the Intervention (Weeks 1-5)
  The EMA items include several investigator designed questions asking participants about the impact of the COVID-19 pandemic, sleep quality, and in-the-moment ratings of anxiety, depression, stress, and loneliness. These are the items that participants will complete every morning. Participants will then be asked to rate in-the-moment anxiety, depression, stress, and loneliness and 3 random points throughout the day. Following week 1, participants will receive prompts about coping with anxiety, stress, uncertainty, and loneliness. Following week 1, participants will also be asked to engage in interoceptive exposure exercises, Intolerance of uncertainty exercises, and loneliness exercises. Participants will be asked to describe their experience of engaging in the exercises using the MetricWire app.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sher L. The impact of the COVID-19 pandemic on suicide rates. QJM. 2020 Oct 1;113(10):707-712. doi: 10.1093/qjmed/hcaa202. PMID 32539153
- [Background] Czeisler ME, Lane RI, Petrosky E, Wiley JF, Christensen A, Njai R, Weaver MD, Robbins R, Facer-Childs ER, Barger LK, Czeisler CA, Howard ME, Rajaratnam SMW. Mental Health, Substance Use, and Suicidal Ideation During the COVID-19 Pandemic - United States, June 24-30, 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 14;69(32):1049-1057. doi: 10.15585/mmwr.mm6932a1. PMID 32790653
- [Background] Mohr DC, Hart SL, Howard I, Julian L, Vella L, Catledge C, Feldman MD. Barriers to psychotherapy among depressed and nondepressed primary care patients. Ann Behav Med. 2006 Dec;32(3):254-8. doi: 10.1207/s15324796abm3203_12. PMID 17107299
- [Background] Brenes GA, Danhauer SC, Lyles MF, Hogan PE, Miller ME. Barriers to Mental Health Treatment in Rural Older Adults. Am J Geriatr Psychiatry. 2015 Nov;23(11):1172-8. doi: 10.1016/j.jagp.2015.06.002. Epub 2015 Jun 17. PMID 26245880
- [Background] Mohr DC, Ho J, Duffecy J, Baron KG, Lehman KA, Jin L, Reifler D. Perceived barriers to psychological treatments and their relationship to depression. J Clin Psychol. 2010 Apr;66(4):394-409. doi: 10.1002/jclp.20659. PMID 20127795
- [Background] DeMartini KS, Carey KB. The role of anxiety sensitivity and drinking motives in predicting alcohol use: a critical review. Clin Psychol Rev. 2011 Feb;31(1):169-77. doi: 10.1016/j.cpr.2010.10.001. Epub 2010 Oct 21. PMID 21074306
- [Background] McClelland H, Evans JJ, Nowland R, Ferguson E, O'Connor RC. Loneliness as a predictor of suicidal ideation and behaviour: a systematic review and meta-analysis of prospective studies. J Affect Disord. 2020 Sep 1;274:880-896. doi: 10.1016/j.jad.2020.05.004. Epub 2020 May 22. PMID 32664029
- [Background] Allan NP, Macatee RJ, Norr AM, Raines AM, Schmidt NB. Relations between common and specific factors of anxiety sensitivity and distress tolerance and fear, distress, and alcohol and substance use disorders. J Anxiety Disord. 2015 Jun;33:81-9. doi: 10.1016/j.janxdis.2015.05.002. Epub 2015 May 21. PMID 26037492
- [Background] Allan NP, Capron DW, Raines AM, Schmidt NB. Unique relations among anxiety sensitivity factors and anxiety, depression, and suicidal ideation. J Anxiety Disord. 2014 Mar;28(2):266-75. doi: 10.1016/j.janxdis.2013.12.004. Epub 2013 Dec 27. PMID 24534564
- [Background] Allan NP, Albanese BJ, Norr AM, Zvolensky MJ, Schmidt NB. Effects of anxiety sensitivity on alcohol problems: evaluating chained mediation through generalized anxiety, depression and drinking motives. Addiction. 2015 Feb;110(2):260-8. doi: 10.1111/add.12739. Epub 2014 Oct 23. PMID 25220033
- [Background] Banducci AN, Bujarski SJ, Bonn-Miller MO, Patel A, Connolly KM. The impact of intolerance of emotional distress and uncertainty on veterans with co-occurring PTSD and substance use disorders. J Anxiety Disord. 2016 Jun;41:73-81. doi: 10.1016/j.janxdis.2016.03.003. Epub 2016 Mar 9. PMID 27004450
- [Background] Allan NP, Boffa JW, Raines AM, Schmidt NB. Intervention related reductions in perceived burdensomeness mediates incidence of suicidal thoughts. J Affect Disord. 2018 Jul;234:282-288. doi: 10.1016/j.jad.2018.02.084. Epub 2018 Feb 27. PMID 29554617
- [Background] Oglesby ME, Allan NP, Schmidt NB. Randomized control trial investigating the efficacy of a computer-based intolerance of uncertainty intervention. Behav Res Ther. 2017 Aug;95:50-57. doi: 10.1016/j.brat.2017.05.007. Epub 2017 May 11. PMID 28531873
- [Background] Raines AM, Allan NP, McGrew SJ, Gooch CV, Wyatt M, Laurel Franklin C, Schmidt NB. A computerized anxiety sensitivity intervention for opioid use disorders: A pilot investigation among veterans. Addict Behav. 2020 May;104:106285. doi: 10.1016/j.addbeh.2019.106285. Epub 2020 Jan 7. PMID 32006788
- [Background] Schmidt NB, Capron DW, Raines AM, Allan NP. Randomized clinical trial evaluating the efficacy of a brief intervention targeting anxiety sensitivity cognitive concerns. J Consult Clin Psychol. 2014 Dec;82(6):1023-33. doi: 10.1037/a0036651. Epub 2014 May 12. PMID 24821096
- [Background] Short NA, Boffa JW, King S, Albanese BJ, Allan NP, Schmidt NB. A randomized clinical trial examining the effects of an anxiety sensitivity intervention on insomnia symptoms: Replication and extension. Behav Res Ther. 2017 Dec;99:108-116. doi: 10.1016/j.brat.2017.09.013. Epub 2017 Oct 5. PMID 29035703
- [Background] Albanese BJ, Macatee RJ, Allan NP, Short NA, Norr AM, Schmidt NB. Interactive Effects of Anxiety Sensitivity and Attentional Control on Posttraumatic Stress in Community and Clinical Populations. Psychiatry. 2018 Spring;81(1):71-84. doi: 10.1080/00332747.2017.1309867. Epub 2018 Mar 22. PMID 29565729
- [Background] Raines AM, Boffa JW, Allan NP, Short NA, Schmidt NB. Hoarding and eating pathology: the mediating role of emotion regulation. Compr Psychiatry. 2015 Feb;57:29-35. doi: 10.1016/j.comppsych.2014.11.005. Epub 2014 Nov 6. PMID 25440599
- [Background] Raines AM, Short NA, Sutton CA, Oglesby ME, Allan NP, Schmidt NB. Obsessive-compulsive symptom dimensions and insomnia: The mediating role of anxiety sensitivity cognitive concerns. Psychiatry Res. 2015 Aug 30;228(3):368-72. doi: 10.1016/j.psychres.2015.05.081. Epub 2015 Jun 28. PMID 26162661
- [Background] Knapp AA, Feldner M, Allan NP, Schmidt NB, Keough ME, Leen-Feldner EW. Test of an Anxiety Sensitivity Amelioration Program for at-risk youth (ASAP-Y). Behav Res Ther. 2020 Mar;126:103544. doi: 10.1016/j.brat.2019.103544. Epub 2020 Jan 2. PMID 31981802
- [Background] Glenn D, Golinelli D, Rose RD, Roy-Byrne P, Stein MB, Sullivan G, Bystritksy A, Sherbourne C, Craske MG. Who gets the most out of cognitive behavioral therapy for anxiety disorders? The role of treatment dose and patient engagement. J Consult Clin Psychol. 2013 Aug;81(4):639-649. doi: 10.1037/a0033403. Epub 2013 Jun 10. PMID 23750465
- [Background] Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker AL, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86. doi: 10.1111/dar.12522. Epub 2017 May 7. PMID 28480521
- [Background] Taylor S, Zvolensky MJ, Cox BJ, Deacon B, Heimberg RG, Ledley DR, Abramowitz JS, Holaway RM, Sandin B, Stewart SH, Coles M, Eng W, Daly ES, Arrindell WA, Bouvard M, Cardenas SJ. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. Psychol Assess. 2007 Jun;19(2):176-88. doi: 10.1037/1040-3590.19.2.176. PMID 17563199
- [Background] Carleton RN, Norton MA, Asmundson GJ. Fearing the unknown: a short version of the Intolerance of Uncertainty Scale. J Anxiety Disord. 2007;21(1):105-17. doi: 10.1016/j.janxdis.2006.03.014. Epub 2006 May 2. PMID 16647833
- [Background] Cyranowski JM, Zill N, Bode R, Butt Z, Kelly MA, Pilkonis PA, Salsman JM, Cella D. Assessing social support, companionship, and distress: National Institute of Health (NIH) Toolbox Adult Social Relationship Scales. Health Psychol. 2013 Mar;32(3):293-301. doi: 10.1037/a0028586. PMID 23437856
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Panchal, N. R. K. C. R. L. C., Kamal, R., Orgera, K., Cox, C., Garfield, R., Hamel, L., ... & Chidambaram, P. (2020). The implications of COVID-19 for mental health and substance use. KFF.
- [Background] NW 1615 L. St, Suite 800Washington, Inquiries D 20036USA202-419-4300 | M-857-8562 | F-419-4372 | M. Demographics of Mobile Device Ownership and Adoption in the United States. Pew Research Center: Internet, Science & Tech. Accessed June 12, 2020. https://www.pewresearch.org/internet/fact-sheet/mobile/
- [Background] Barlow DH, Craske MG. Mastery of Your Anxiety and Panic. Oxford University Press; 2006.
- [Background] Cully JA, Teten AL. A therapist's guide to brief cognitive behavioral therapy. Houst Dep Veterans Aff South Cent MIRECC. Published online 2008.
- [Background] Thase ME, Callan JA. The role of homework in cognitive behavior therapy of depression. J Psychother Integr. 2006;16(2):162-177. doi:10.1037/1053-0479.16.2.162
- [Background] Sheehan D, Janavs J, Baker R, Sheehan KH, Knapp E, Sheehan M. Mini International Neuropsychiatric Interview-Version 7.0. 0 DSM-5. 2014.; 2015.
- [Background] Kinser PA, Robins JL. Control group design: enhancing rigor in research of mind-body therapies for depression. Evid Based Complement Alternat Med. 2013;2013:140467. doi: 10.1155/2013/140467. Epub 2013 Apr 7. PMID 23662111